CLINICAL TRIAL: NCT01272284
Title: The Altis® Single Incision Sling System for Female Stress Urinary Incontinence Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP006SU
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Stress Urinary Incontinence
Keywords: Female; Stress urinary incontinence; Mini sling; Single incision sling; Urinary incontinence; Mixed urinary incontinence; Additional relevant MESH terms:; Stress; Urinary Incontinence, Stress; Pathological Processes; Urination Disorders; Urological Disorders; Urological Manifestations; Signs and Symptoms
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Pathologic Processes; Urination Disorders; Urologic Diseases; Urological Manifestations; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altis® SIS (Other): Subjects enrolled with Altis® SIS
  Interventions: Device: Altis® Single Incision Sling System (SIS)

INTERVENTIONS:
Device: Altis® Single Incision Sling System (SIS) — The Altis® SIS is a permanently implantable synthetic sling for females placed at the mid-urethra to provide a scaffold for tissue in-growth and support for stress urinary incontinence.

SUMMARY:
An international, multi-center, single arm, prospective clinical study designed to assess the safety and efficacy of the Coloplast Altis single incision sling system for females with stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
An international, multi-center, single arm, prospective clinical study designed to assess the safety and efficacy of the Coloplast Altis single incision sling system for females with stress urinary incontinence (SUI). Primary Objective: Improvement in continence measured by 24 hour pad weight test with at least a 50% reduction in weight from baseline at 6 months. Secondary Objectives: Cough stress test results at 6 months; Subject QoL as measured by validated questionnaires: PGI-I, improvements in UDI-6 and IIQ-7 scores from baseline at 6 months, 3 day voiding diary improvement from baseline at 6 months; Device and procedure related adverse events. Brief Entrance Criteria: Adult female with confirmed SUI through cough stress test or urodynamics; Failed two non-invasive incontinence therapies; No prior surgical SUI treatment; No prolapse POP-Q Stage 2 or higher; No concurrent pelvic floor procedure; No urge predominant incontinence; No incontinence due to neurological disorder/disease; No PVR > 100cc; and, No contraindication to the surgical procedure. Study visits will take place at baseline, implant/hospitalization, 3 months, 6 months, 1 year, and 2 years post operatively. This study will enroll up to 113 subjects at up to 17 investigative sites in the US and Internationally.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female at least 18 years of age
* Subject is able and willing to complete all procedures and follow-up visits indicated in this protocol
* Subject has confirmed stress urinary incontinence (SUI) through cough stress test or urodynamics
* The subject has failed two non-invasive incontinence therapies (such as Kegel exercise, behavior modification, pad use, biofeedback, etc) for >6 months

Exclusion Criteria:

* Subject has an active urogenital infection or active skin infection in region of surgery
* Subject has confirmed Pelvic Organ Prolapse (POP) of Stage 2 or higher as determined by POP-Q prolapse grading
* Subject is having a concomitant pelvic floor procedure
* Subject has incontinence due to neurogenic causes (e.g. multiple sclerosis, spinal cord/brain injury, cerebrovascular accident, detrusor-external sphincter dyssynergia, Parkinson's disease, or similar conditions)
* Subject had a prior surgical SUI treatment
* Subject has undergone radiation or brachy therapy to treat pelvic cancer
* Subject has urge predominant incontinence
* Subject has an atonic bladder or a post void residual (PVR) consistently about 100cc
* Subject is pregnant and/or is planning to get pregnant in the future
* Subject has a contraindication to the surgical procedure or the Altis Instructions For Use (IFU)
* Subject is enrolled in a concurrent clinical trial of any treatment (drug or device) that could affect continence function without the sponsor's approval

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Kocjancic, MD, Principal Investigator — University of Chicago, Chicago, IL, United States
Locations (17):
- United States (16):
  - Tri Valley Urology, Murrieta, California
  - Urology Specialists, LLC, Hialeah, Florida
  - Atlanta Medial Research Institute, Alpharetta, Georgia
  - Rosemark Womencare Specialist, Idaho Falls, Idaho
  - University of Illinois at Chicago - Department of Urology, Chicago, Illinois
  - Illinois Urogynecology, LTD, Oak Lawn, Illinois
  - Female Pelvic Medicine & Urogynecology Institute of Michigan, Grand Rapids, Michigan
  - Bellevue ObGyn, Bellevue, Nebraska
  - Delaware Valley Urology, Voorhees Township, New Jersey
  - Carolina Urology Partners, Gastonia, North Carolina
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Greenville Hospital System, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - The Group for Women, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Johnston Willis Medical Center, Richmond, Virginia
- CHUS Hopital Fleurimont, Sherbrooke, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with documented stress urinary incontinence (SUI) who met enrollment criteria
Groups:
- Altis® SIS: Participants implanted with Altis® Single Incision Sling
Period: 3-month Follow-up Visit
Arm/Group | Altis® SIS
Started | 113
Completed | 112
Not Completed | 1
Period: 6-month Follow-up Visit
Arm/Group | Altis® SIS
Started | 112
Completed | 109
Not Completed | 3
Period: 12-month Follow-up Visit
Arm/Group | Altis® SIS
Started | 109
Completed | 105
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Altis® SIS
Number analyzed (Participants) | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 86
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 93
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 50% Reduction in 24-hour Pad Weight From Baseline to 6 Months
Description: Primary endpoint defined as at least a 50% reduction in 24-hour pad weight from baseline to 6 months (including dry as defined as a pad weight of less than 1.3 grams during the 6-month test), in which the percent of subjects with at least 50% reduction in 24-hour pad weight is compared to a performance goal of 50%.
Time Frame: 6 months (compared to baseline)
Population: Analysis was per protocol. 109 subjects were eligible for 6-month follow-up. 6 subjects missed either the visit or the pad weight test.
Measure: Number; unit: percentage of participants
Groups:
- Altis SIS®: Participants implanted with Altis® Single Incision Sling
Arm/Group | Altis SIS®
Number analyzed (Participants) | 103
percentage of participants | 85.4
Statistical Analysis 1: Comparison: Altis SIS®; The final significance level is 0.04191 accounting for one interim analysis conducted at 80% of final information, thus a 95.81% Confidence Limit (CL) was used; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Proportion successful = 85.4, 95.81% CI 1-sided [lower limit 78.1]

2. Secondary Outcome: Percentage of Participants With Negative Cough Stress Test at 6 Months
Description: Endpoint defined as a negative result at 6 months, as measured by the Cough Stress Test (CST), in which the percent of subjects with a negative CST is compared to a performance goal of 66%.
  The cough stress test was completed with the subject in the lithotomy and standing positions, filling bladder to maximum capacity with normal saline. The subject was then asked to cough 10 times and any leakage from the urethra was considered a positive test.
Time Frame: 6 months
Population: 109 subjects were eligible for 6-month follow-up. 6 subjects missed either the visit or the cough stress test.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 103
percentage of participants | 92.2

3. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in Incontinence Via 3-Day Voiding Diary From Baseline to 6 Months
Description: Endpoint defined as at least a 50% improvement from baseline to 6-months, as measured by 3-Day Voiding Diary, in which the percent of subjects with at least a 50% improvement from baseline to 6 months is compared to a performance goal of 50%.
  Subjects completed a 3-Day Voiding Diary of controlled urinations and the number and amount of leaks experienced.
Time Frame: 6 months (compared to baseline)
Population: 109 subjects were eligible for 6-month follow-up. 17 subjects either missed the visit or did not complete the 3-Day Voiding Diary.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 92
percentage of participants | 88

4. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in UDI-6 Score From Baseline to 6 Months
Description: Endpoint defined as at least a 50% improvement from baseline to 6 months, as measured by validated Urinary Distress Inventory Short Form (UDI-6), in which the percent of subjects with at least a 50% improvement from baseline to 6 months is compared to a performance goal of 50%.
Time Frame: 6 months (compared to baseline)
Population: 109 subjects were eligible for 6-month follow-up. 4 subjects either missed the visit or did not complete the Urinary Distress Inventory.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 105
percentage of participants | 88.6

5. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in IIQ-7 From Baseline to 6 Months
Description: Endpoint defined as at least a 50% improvement from baseline to 6 months, as measured by validated Incontinence Impact Questionnaire Short Form (IIQ-7), in which the percent of subjects with at least a 50% improvement from baseline to 6 months is compared to a performance goal of 50%.
Time Frame: 6 months (compared to baseline)
Population: 109 subjects were eligible for 6-month follow-up. 5 subjects either missed the visit or did not complete the Incontinence Impact Questionnaire.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 104
percentage of participants | 93.3

6. Secondary Outcome: Percentage of Patients Responding "Very Much Better" or "Much Better" on PGI-I at 6 Months
Description: Success defined as a response of "Very Much Better" or "Much Better" at 6 months, as measured by validated Patient Global Impression of Improvement (PGI-I).
Time Frame: 6 months
Population: 109 subjects were eligible for 6-month follow-up. 4 subjects either missed the visit or did not complete the PGI-I.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 105
percentage of participants | 87.6

7. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in 24-hour Pad Weight From Baseline to 12 Months
Description: Success is defined as at least a 50% reduction in 24-hour pad weight from baseline to 12 months using the 24 hour pad weight test.
Time Frame: 12 months (compared to baseline)
Population: 105 subjects were eligible for 12-month follow-up. 4 subjects missed either the visit or the pad weight test.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 101
percentage of participants | 90.1

8. Secondary Outcome: Percentage of Participants With Negative Cough Stress Test at 12 Months
Description: Success defined as a negative result at 12 months, as measured by the Cough Stress Test (CST).
  The cough stress test was completed with the subject in the lithotomy and standing positions, filling bladder to maximum capacity with normal saline. The subject was then asked to cough 10 times and any leakage from the urethra was considered a positive test.
Time Frame: 12 months (compared to baseline)
Population: 105 subjects were eligible for 12-month follow-up. 4 subjects missed either the visit or the cough stress test.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 101
percentage of participants | 90.1

9. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in UDI-6 Score From Baseline to 12 Months
Description: Success defined as at least a 50% improvement from baseline to 12 months, as measured by validated Urinary Distress Inventory Short Form (UDI-6)
Time Frame: 12 months (compared to baseline)
Population: 105 subjects were eligible for 12-month follow-up. 2 subjects either missed the visit or did not complete the UDI-6.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 103
percentage of participants | 89.3

10. Secondary Outcome: Percentage of Participants With at Least 50% Improvement in IIQ-7 From Baseline to 12 Months
Description: Success defined as at least a 50% improvement from baseline to 12 months, as measured by validated Incontinence Impact Questionnaire Short Form (IIQ-7)
Time Frame: 12 months (compared to baseline)
Population: 105 subjects were eligible for 12-month follow-up. 2 subjects either missed the visit or did not complete the IIQ-7.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 103
percentage of participants | 90.3

11. Secondary Outcome: Percentage of Patients Responding "Very Much Better" or "Much Better" on PGI-I at 12 Months
Description: Success defined as a response of "Very Much Better" or "Much Better" at 12 months, as measured by validated Patient Global Impression of Improvement (PGI-I).
Time Frame: 12 months
Population: 105 subjects were eligible for 12-month follow-up. 2 subjects either missed the visit or did not complete the PGI-I.
Measure: Number; unit: percentage of participants
Arm/Group | Altis® SIS
Number analyzed (Participants) | 103
percentage of participants | 89.3

ADVERSE EVENTS:
Arm/Group | Altis® SIS
Serious Adverse Events (participants affected / at risk) | 3/113
Other Adverse Events (participants affected / at risk) | 9/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Altis® SIS (N=113)
Hematoma (Surgical and medical procedures) | 1 (1) — Pelvic hematoma, resolved spontaneously in hospital
Mesh extrusion (Surgical and medical procedures) | 1 (1) — Subject underwent surgical revision due to symptoms
Mesh extrusion (Surgical and medical procedures) | 1 (1) — Classified as serious adverse event (SAE) due to subject withdrawal from study prior to further follow-up data collection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Altis® SIS (N=113)
Non-pelvic pain (Surgical and medical procedures) | 9 (9) — Procedure-related non-pelvic pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less